CLINICAL TRIAL: NCT01641900
Title: Sleep-dependent Memory Processing in Schizophrenia
Brief Title: Effects of Eszopiclone on Sleep and Memory in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Mclean Hospital (Other)
Responsible Party: Principal Investigator, Dara S. Manoach, PhD, Professor of Psychology, Dept. of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01MH092638 (NIH)
Record Dates: First submitted 2012-01-25; First posted 2012-07-17 (Estimated); Results first posted 2017-05-16 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Schizophrenia
Keywords: sleep; memory; schizophrenia; eszopiclone
MeSH Terms: conditions — Schizophrenia | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Schizophrenia (Experimental): Outpatients with a Structural Clinical Interview confirmed DSM-IV diagnosis of schizophrenia.
  All participants receive two interventions: 3 mg eszopiclone and Placebo Intervention conditions are separated by 1 week.
  Interventions: Drug: eszopiclone; Drug: placebo
- Healthy Controls (Experimental): Adult participants screened to exclude a personal history of mental illness, family history of schizophrenia spectrum disorder, and psychoactive medication use. All participants receive two interventions: 3 mg eszopiclone and Placebo Intervention conditions are separated by 1 week.
  Interventions: Drug: eszopiclone; Drug: placebo

INTERVENTIONS:
Drug: eszopiclone — 3 mg of eszopiclone for two consecutive nights (Baseline Night and Experimental Night). Sleep spindle density (primary outcome) is measured for both nights. Memory consolidation (secondary outcome) is measured over Experimental Night.
  Other Names: Lunesta
Drug: placebo — placebo capsule for two consecutive nights. (Baseline Night and Experimental Night). Sleep spindle density (primary outcome) is measured for both nights. Memory consolidation (secondary outcome) is measured over Experimental Night.

SUMMARY:
The investigators will test the hypothesis that the sleep medication, eszopiclone, can normalize brain activity during sleep and improve memory in patients with schizophrenia. The investigators will do this by measuring sleep and memory performance on two conditions separated by one week: taking 3 mg of eszopiclone and taking placebo. The investigators will study healthy subjects and chronic, medicated outpatients with schizophrenia.

DETAILED DESCRIPTION:
Sleep spindles, a defining oscillation of stage 2 non-rapid eye movement sleep (N2), are strongly linked to memory and IQ in healthy individuals. Schizophrenia is characterized by a spindle deficit that correlates with deficient sleep-dependent memory consolidation, symptom severity, IQ and executive function. In a small pilot study of schizophrenia patients, eszopiclone , significantly increased sleep spindles but its effect on memory was not significant. Here, in a larger double-blind, placebo-controlled, cross-over design study, we investigated whether eszopiclone can both increase spindle density and improve memory consolidation. Chronic, medicated schizophrenia outpatients and demographically-matched healthy control participants were randomly assigned to receive either placebo first or 3mg of eszopiclone first for two consecutive nights with high density polysomnography. Placebo and eszopiclone visits were one week apart. Participants were trained on the Motor Sequence Task (MST) at bedtime of the second night of each visit and tested the following morning to probe sleep-dependent motor memory consolidation.

ELIGIBILITY:
Inclusion Criteria:

* clinically stable outpatients with schizophrenia,
* proficient in English,
* able to give informed consent,
* maintained on a stable dose of atypical antipsychotic medications for at least 6 weeks prior to enrollment.
* healthy Control participants matched as a group to the patients for age, sex, and parental socioeconomic status.

Exclusion Criteria:

* Substance abuse or dependence within the past six months;
* other chronic medical conditions that affect sleep; (- pregnancy/breast feeding;
* hepatic impairment;
* treatment with inhibitors or inducers of CYP 3A4 or 2E1 enzymes (which metabolize eszopiclone);
* a history of head injury resulting in prolonged loss of consciousness or other neurological sequelae; (- mental retardation; (- a diagnosed sleep disorder other than insomnia,
* neurological disorder; sleep disorder, other than insomnia, identified in a clinical sleep evaluation.

Patients on conventional agents, benzodiazepines, or other sleep agents will be excluded. Potential controls will be excluded for a personal history of mental illness, a family history of schizophrenia spectrum disorder or psychosis, and treatment with medications known to affect sleep or cognition.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2012-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dara S Manoach, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD data.

RESULTS

PARTICIPANT FLOW:
Groups:
- Group: Schizophrenia: Outpatients with a Structural Clinical Interview confirmed DSM-IV diagnosis of schizophrenia. Participants completed both the Drug and Placebo arms.
- Group: Healthy Controls: Adult participants screened to exclude a personal history of mental illness, family history of schizophrenia spectrum disorder, and psychoactive medication use. Participants completed both the Drug and Placebo arms.
Period: Overall Study
Arm/Group | Group: Schizophrenia | Group: Healthy Controls
Started | 28 | 31
Completed Placebo Intervention | 27 (n=1,assigned to placebo intervention first, completed the session and dropped out of the study.) | 29 (n=2,both assigned to placebo intervention first, completed the session and dropped out of the study.)
Completed Drug Intervention | 26 (n=1,assigned to drug intervention first, completed the session and dropped out of the study.) | 29
Completed | 26 | 29
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Population: All participants completed both the Drug and Placebo arms
Groups:
- Total: Total of all reporting groups
Arm/Group | Group: Schizophrenia | Group: Healthy Controls | Total
Number analyzed (Participants) | 26 | 29 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 29 | 55
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (7.5) | 30.1 (6.2) | 31.13 (6.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 21 | 21 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 19 | 19 | 38
  Unknown or Not Reported | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 0 | 6
  White | 12 | 17 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 9 | 14
Region of Enrollment [Number; unit: participants]
  United States | 26 | 29 | 55

OUTCOME MEASURES:

1. Primary Outcome: Sleep Spindle Density
Description: This measure is averaged for Baseline and Experimental nights. Sleep spindle density (number/minute) for non-Rapid Eye Movement Stage 2 sleep (N2) detected at channel Cz based on polysomnographic recordings.
Time Frame: Spindles will be averaged for the Baseline (Night 1) and Experimental Nights (Night 2)
Measure: Mean (Standard Deviation); unit: Sleep spindle density (number/minutes)
Arm/Group | Group: Schizophrenia | Group: Healthy Controls
Number analyzed (Participants) | 26 | 29
Sleep spindle density (number/minutes)
  Placebo (placebo capsule) | 2.02 (0.44) | 2.13 (0.51)
  Drug (3mg eszopiclone) | 2.25 (0.41) | 2.44 (0.44)

2. Secondary Outcome: Motor Procedural Memory Performance
Description: Overnight performance improvement on the finger tapping motor sequence task (MST).The MST involves pressing four numerically labeled keys on a standard keyboard with the fingers of the left hand, repeating a 5 digit sequence as quickly and accurately as possible for 12 trials at 30 seconds each separated by 30 sec rest periods. Different sequences were employed for the Placebo and Drug visits in a counter-balanced order. MST performance is measured as the number of correctly typed sequences in each trial. The primary outcome measure is overnight improvement calculated as the percent increase in average of correct sequences from the last three training trials to the average of first three test trials. Since the outcome measure is calculated as percent improvement from training to test for each participant, there is no highest or lowest possible score.
Time Frame: Experimental Night (Night 2)
Measure: Mean (Standard Deviation); unit: percentage of improvement on MST perform
Arm/Group | Group: Schizophrenia | Group: Healthy Controls
Number analyzed (Participants) | 26 | 29
percentage of improvement on MST perform
  Placebo (Placebo capsule) | 13.35 (15.62) | 15.1 (12.22)
  Drug (3mg eszopiclone) | 9.69 (17.53) | 16.69 (17.14)

ADVERSE EVENTS:
Time Frame: through study completion
Groups:
- Placebo With Schizophrenia: Outpatients with a Structural Clinical Interview confirmed DSM-IV diagnosis of schizophrenia. Participants who completed Placebo Intervention.
- Placebo Healthy Controls: Adult participants screened to exclude a personal history of mental illness, family history of schizophrenia spectrum disorder, and psychoactive medication use.Participants who completed Placebo Intervention.
- 3mg Eszopiclone With Schizophrenia: Outpatients with a Structural Clinical Interview confirmed DSM-IV diagnosis of schizophrenia. Participants who completed Drug Intervention.
- 3mg Eszopiclone Healthy Controls: Adult participants screened to exclude a personal history of mental illness, family history of schizophrenia spectrum disorder, and psychoactive medication use.Participants who completed Drug Intervention.
Arm/Group | Placebo With Schizophrenia | Placebo Healthy Controls | 3mg Eszopiclone With Schizophrenia | 3mg Eszopiclone Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/31 | 0/28 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/31 | 0/28 | 0/31
Other Adverse Events (participants affected / at risk) | 0/28 | 0/31 | 0/28 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No